CLINICAL TRIAL: NCT01191281
Title: Improving Food Security and Nutrition to Promote ART Adherence in Latin America
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Homero Martinez, Senior Social Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRANT00395147; R34MH084675-02 (NIH)
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Medication Adherence
Keywords: food habits; nutrition requirements; antiretroviral therapy
MeSH Terms: conditions — Medication Adherence; Feeding Behavior | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet/nutrition counsel+food aid (Experimental): Intervention. Patients enrolled in the intervention group will receive a multi-component intervention that includes dietary and nutritional counseling and food assistance (food aid basket)
  Interventions: Behavioral: Diet/nutrition counsel+food aid
- dietary/nutritional counseling (Active Comparator): Patients enrolled in the comparison arm will receive dietary and nutrition counseling designed to help them meet their nutrition needs, based on foods which are locally available, culturally acceptable and within their budget.
  Interventions: Other: Dietary/nutrition counsel

INTERVENTIONS:
Behavioral: Diet/nutrition counsel+food aid — Patients enrolled in the experimental arm will receive dietary and nutritional assistance plus a food aid basket, specifically tailored to meet the nutritional needs of the target population.
  Arms: Diet/nutrition counsel+food aid
Other: Dietary/nutrition counsel — Patients enrolled in the active comparison arm will receive dietary and nutrition counseling designed to help them meet their nutrition needs, based on foods which are locally available, culturally acceptable and within their budget.
  Arms: dietary/nutritional counseling

SUMMARY:
The purpose of this three-year study is to develop, implement, and pilot test a culturally appropriate, multi-component nutrition intervention for people living with HIV and food insecurity in Honduras, which is among the Latin America nations with the highest HIV prevalence rates. The investigators specific aims are to:

1. Explore the relationships between food security, nutrition, and HIV treatment access, utilization, and adherence, and examine key mediators and moderators of these relationships.
2. Develop a multi-component nutrition intervention to address food insecurity among Honduran HIV+ individuals and their families.
3. Evaluate the preliminary effectiveness of the intervention on (1) food security and nutritional status; (2) HIV care retention (clinic attendance), uptake of ART when recommended, and ART adherence; and (3) clinical outcomes (CD4 count, ART side effects, and opportunistic infections).
4. Examine key mediators and moderators of the intervention effects from among characteristics of the patient, household, and contextual setting.

DETAILED DESCRIPTION:
The project will be conducted in two phases. Phase 1 involves qualitative, formative research methods to (1) gain understanding of availability and cost of the local foods and the regular diet, (2) evaluate the level of food security among people living with HIV, including intra-household food distribution patterns, and assess the nutritional status of HIV affected individuals, and (3) examine the role that food security and nutrition play in HIV treatment access, utilization and adherence. Phase 2 consists of developing and pilot-testing a multi-component nutrition intervention through a randomized, controlled trial conducted at 4 HIV clinics in Honduras, with two clinics randomly assigned to receive the intervention and two clinics to serve as the comparison group. Patients at each of the 4 sites will receive nutrition counseling, following the guidelines currently proposed by the World Health Organization (WHO) as the standard of care for HIV-infected individuals. In addition, clients at the intervention sites will receive food assistance in the form of a food-aid basket, designed ad hoc to address their macro and micronutrient needs.

ELIGIBILITY:
Inclusion Criteria:

* Registered at the clinic
* Age 18 or older
* If not on ART, CD4 < 350*
* Living in the area for the past year.

Exclusion Criteria:

* Deterioration of clinical status such that requires diet or nutrition therapy
* Cannot understand or speak Spanish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ART uptake and adherence | Monthly during 12 of follow-up
Nutritional status | Monthly during 12 months of follow-up
  Nutritional status will be assess by anthropometry every month during follow-up

SECONDARY OUTCOMES:
HIV clinical outcomes | At 6 and 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Homero Martinez, PhD, Principal Investigator — RAND
Locations (1):
- RAND Corporation, Santa Monica, California, United States